CLINICAL TRIAL: NCT06732479
Title: Effectiveness of Behavioural Skills Training (BST) on Knowledge of Sexual Abuse and Resistance Ability Among Children with Intellectual Disabilities: a Randomized Controlled Trial
Brief Title: Behavioural Skills Training (BST) for Teaching Sexual Abuse Prevention Skills for Children with Intellectual Disabilities
Acronym: BST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Canberra (Other)
Collaborators: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, Natasha Jojo, Assistant Professor, University of Canberra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIMHANS/DO/101ST IEC/2015; NIMH:A&E/C:Ph.D(Nsg):2014-16:N (Other: National Institute of Mental Health and Neuro Sciences, Bangalore)
Record Dates: First submitted 2024-12-08; First posted 2024-12-13 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Intellectual Disability, Mild to Moderate; Sexual Abuse
Keywords: Behavioural Skills Training; children with intellectual disabilities; Sexual abuse prevention; sexual abuse and resistance ability
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Intervention Model Description: Participants were systematically selected using a stratified random sampling approach. The schools were first categorised into three strata based on the number of enrolled children: those with more than 100 children, those between 25 and 100 children, and those with fewer than 25 children. Schools were randomly chosen from each stratum. Two schools with more than 100 children were randomly selected, one designated as the experimental group and the other as the control group. Six schools in the 25 to 100 children were randomly chosen and equally divided into experimental and control groups. Similarly, in the stratum of schools with less than 25 children, four schools were randomly selected and equally split into experimental and control groups. It is important to note that all participants who met the predetermined selection criteria within each selected school for specific purposes were invited to participate in the study, ensuring a comprehensive and representative sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group: Treatment as usual (TAU) (No Intervention): These included general safety tips, and the detailed instructions taught to children by teachers in special school during academic programme. As part of the curriculum, teachers taught children about safe touch and unsafe touch and instructed children to say "No" to unsafe touches. Teachers mainly focused on inappropriate touches and the main mode of instruction was lecturing.
- Behavioral skill Training (BST) (Experimental): The Behavioural Skill Training (BST) was developed by modifying the Body Safety Training programme developed by Dr.Sandy.K.Wurtele.The Module was organized under 10 lessons. Each lesson was taught through stories, and each story had a picture that goes along with it. Children were taught first about the general safety (poison safety, fire safety, pedestrian safety, and vehicle safety) as a way of establishing rapport, and then moved to body safety rules (stranger safety, concept of private parts, appropriate and inappropriate touches, self-protection skills). Appropriate and inappropriate situations were presented using video and training was given to children on how to respond appropriately to each situation using role play. The Module was delivered over a period of one month, three sessions per week.
  Interventions: Behavioral: Behavioural Skill Training Programme

INTERVENTIONS:
Behavioral: Behavioural Skill Training Programme — BST was administered in 3 sessions in a week on alternate days, each session lasting for an hour. Training was given in small groups consisting of 4-6 members. Parents were involved as co-therapists, and observed the training given by the researcher and practiced it at home with their children.
  The training was carried out through the following steps:
  1. Instruction- Involved teaching the location of private parts, difference between appropriate and inappropriate touch, safe and unsafe secrets, sexuality, self-protection skills (saying NO, move from situation, tell trusted person, report the person and situation.
  2. Modelling- researcher, modelled, correct responses, and instructed to act in the unsafe situation using role play. Situations were presented using video.
  3. Rehearsal-researcher presented situations using video and instructed to rehearse the skills until able to demonstrate the skill independently
  Arms: Behavioral skill Training (BST)

SUMMARY:
The main goal of the study was to see if Behavioural Skills Training (BST) could improve knowledge about sexual abuse and the ability to resist it among children with intellectual disabilities. This study also evaluated any negative effects of the programme on children with intellectual disabilities. There were two groups, one group received a training programme which was delivered as three one-hour sessions in a week over 12 weeks. The Behavioral Skills Training (BST) module was structured into ten lessons, each conveyed through engaging stories and corresponding illustrations. The training commenced with teaching children general safety topics such as poison, fire, pedestrian, and vehicle safety. This served as an initial step to establish comfort.

Subsequently, the module transitioned to imparting knowledge on body safety rules. This included educating children on stranger safety and private parts, understanding appropriate and inappropriate touches, and teaching them self-protection skills. Videos were used to show appropriate and inappropriate situations effectively, and training sessions involved role-playing scenarios. Another group received the usual sex education offered by teachers at school. After completing training students were assessed for their knowledge regarding sexual abuse and their self-protection skills (ability to say no, remove themselves from the situation, identify a person to whom the incident can be reported and report the incident and identify the offender. This was assessed based on the situations presented in a video. Children were tested one week after the training, at one-month, three-month and six-month intervals to see whether they could retain the information and skill. Their knowledge and self-protection skills improved after attending the programme and it was retained for six months. Participation in the programme did not cause any negative effects among children with intellectual disabilities.

DETAILED DESCRIPTION:
Sexual abuse of children with intellectual disabilities is a global concern. Rate of sexual abuse among children with intellectual disabilities is 2-4 times the rate in general population. Thirty-nine to 83% of girls and 16%- 32% of boys with Intellectual Disability typically experience sexual abuse by the time they reach the age of 18. There is a need for personal safety programs as one of the multiple approaches to reduce the risk of child sexual abuse. In order to protect themselves against abuse, children with intellectual disability must have the skills to independently recognise potentially abusive situations and respond appropriately. Even though some of the abuse prevention programmes are widely used, the effectiveness of these is not established. The aim of the study was to assess the effectiveness of a Behavioural Skills Training on knowledge of sexual abuse and resistance ability among children with Intellectual Disability.

Sample size calculation for this study was conducted using power analysis, based on the variance from the pilot study. Considering a statistical power of 80% and a significance level set at 5%, 134 children were initially recruited for the study. However, upon concluding the six months, data was available to only 120 subjects. Among these, 60 children received the intervention ( experimental group), while the remaining 60 received Treatment as Usual (the control group).

This study developed a Video based Behavioural Skill Training programme for training children with intellectual disabilities for improving their knowledge regarding sexual abuse and resistance ability against sexual abuse and tested its effectiveness. The study involved children initially watching video presentations depicting appropriate and inappropriate situations and the ideal responses for each scenario. Subsequently, the children engaged in role-playing exercises, where a researcher assumed the roles of a perpetrator, doctor, or nurse. At the same time, parents who participated as co-therapists in the study played their parents' part in the role play. Following each enactment of inappropriate situations, the children were instructed to approach their parents and report the individual's identity and the incident. This role-playing process was reiterated until the children had comprehensively learned the appropriate responses.

The effectiveness of the study was evaluated based on the change in the knowledge scores and resistance ability scores. A randomized controlled design with longitudinal measurement of outcomes was adopted to evaluate the effectiveness of BST on Knowledge of Sexual Abuse and Resistance Ability. Screening for all the children was done in each selected special schools based on the inclusion and exclusion criteria. All subjects who met the criteria were selected for the study.

The children and parents involved in the study were clearly informed about its purpose and objectives. Written informed consent was obtained from the parents, and an attempt was made to obtain assent from the children. Forty-two percent of the children were able to provide signed assent. Participants were assured that the information they provided would remain confidential. It was also ensured that the BST would not interfere with the children's regular school schedules. The investigator closely monitored the children and their parents during the intervention to address any potential adverse effects.

At the outset of our research project, we initiated meetings with parents and children to establish mutual understanding and rapport. The teachers played a crucial role in interactions with the parents and children. They helped establish contact with the parents and took on the role of introducing us to both the parents and the children. Their support and involvement were instrumental in creating a welcoming and cooperative atmosphere for our research endeavours. During these meetings, we encouraged parents and children to ask any questions they had about the research. This open and transparent dialogue was a valuable foundation for collaborative efforts and ensured that all parties involved were well-informed and comfortable with the research process.

The introduction to the children was facilitated by the class teacher, allowing us to interact with them within the classroom setting before conducting interviews. This preliminary interaction reduced any sense of unfamiliarity or apprehension among the children. Prior to commencing the interviews, we obtained assent from each child. We informed them that we would ask questions about personal safety and protecting themselves in various situations.

Each child was individually interviewed in an open classroom or library, ensuring a comfortable and non-intimidating environment. The administration sequence first involved conducting the Personal Safety Questionnaire (PSQ) and the video-enhanced 'What If Situation Test' (WIST). Both assessments were administered orally, with responses recorded on paper-based tools. The sessions were conducted in small groups, typically consisting of children, within classroom settings, library halls, or auditoriums. It is essential to note that the child's parents also actively participated in these training sessions and were encouraged to reinforce the training at home. Each training session had a duration of approximately 1 hour.

To analyse the data, verbatim interview responses were coded, with scores assigned for each question or item. This systematic approach allowed for a comprehensive assessment of the children's understanding of personal safety and their ability to respond effectively to various situations.

After the study's completion, the BST was also provided to the control group. Subjects in the experimental and control group was assessed for their knowledge and resistance ability before the intervention and post assessment was done after the intervention. Descriptive statistics were applied for the baseline data. Descriptive statistics includes frequency distributions, mean and median for the central tendency and range and standard deviation. Chi square was done to find the association between the categorical variables. To assess the effectiveness of the intervention program, Mann Whitney U was done to compare the outcome measures between the experimental and control group All the analysis was performed in IBM SPSS statistics 22 and a p-level of <0.05 was considered as statistically significant. Mean age (in years) of the total sample (n=120) was 15.6 ±2.6 and it was 15.3 ± 2.7 in experimental group (n=60) and 15.9 ± 2.5 in control group (n=60). In the sample 59.2% of the children belonged to the category of mild intellectual disabilities and rest were with moderate intellectual disabilities.

The BST was found to be effective in increasing knowledge (P<0.01) regarding sexual abuse and resistance ability (P<0.01) against sexual abuse among children with mild or moderate disabilities.

ELIGIBILITY:
Children

Inclusion criteria:

* Children with mild and moderate Intellectual Disability as per Diagnostic and Statistical manual (DSM) V, and as determined by the assessment of qualified educational psychologists prior to the admission to the special schools.
* Age 10-18 years
* Those children whose parents are available during the period of study
* Children with verbal ability which would allow them to participate in the study

Exclusion criteria:

* Children who cannot speak Malayalam/English
* Presence of active symptoms of co morbid psychiatric illness

Parent

Inclusion criteria

* Parents (either mother or father) who are willing to participate as co therapists.
* Parents staying with the child for at least for one year and are the primary care givers of the child. Exclusion criteria
* Parents who cannot speak Malayalam/ English
* Parents who are not willing to participate in the one month,3 month and 6 month follow ups.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2017-03-11 (Actual); Study Completion 2017-03-11 (Actual)

PRIMARY OUTCOMES:
Personal Safety Questionnaire | pre intervention and one week, one month, 3 month and 6 months after the intervention
  Designed to evaluate knowledge regarding sexual abuse, this questionnaire consists of 11 items related to personal safety. Participants respond with "yes," "no," or "I do not know" to these items, and scores can range from 0 to 11; a higher score indicates a more comprehensive understanding of sexual abuse. The score range spans from 0 to 11, with an average score of 5.5. Personal Safety Questionnaire (PSQ) demonstrates strong test-retest reliability (r = 0.77) and internal consistency (Cronbach's α = 0.78).
Video supplemented 'what if' situation test | pre intervention and one week, one month, 3 month and 6 months after the intervention
  This test assesses the participant's ability to differentiate appropriate from inappropriate sexual advances and their understanding of hypothetical abusive situations. It includes two practice trials and six brief vignettes. Three vignettes describe appropriate requests for touch, while the other three depict inappropriate requests. The 'What If Situation Test' generates three scale scores: 1) Appropriate request recognition (score range: 0-3), 2) Inappropriate request recognition (score range: 0-3), 3) Total score, which measures knowledge of self-protection skills (score range: 0-24). The total score comprises four specific skill scores that represent the participant's verbal reports on their ability to 1) Refuse advances using appropriate, assertive, and persistent verbal responses (say), 2) Remove themselves from the situation (do), 3) Identify a person to whom the incident can be reported (tell) 4) Report the incident and identify the offender.

SECONDARY OUTCOMES:
Side effects measure | pre intervention and one week, one month, 3 month and 6 months after the intervention
  The 12-item fear assessment thermometer scale assessesparticipants' fear of various objects, people and situations. Participants' fear is rated by moving a simulated mercury column from 1 (not at all afraid) to 7 (very much afraid)on a card board representation of a thermometer. Scores ranged from 12 to 84.
  After the pilot study, this scale was modified with the permission of the original author, since the children had difficulty to differentiate seven categories, and hence categories were changed to very much afraid (3), slightly afraid (2), not at all afraid (1). The revised scores range from 12 to 36.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Natasha Jojo, PhD, Principal Investigator — University of Canberra

IPD SHARING:
Plan to Share IPD: No
This will not be shared to protect the confidentiality and privacy of the participants

REFERENCES:
- [Background] Schaafsma D, Kok G, Stoffelen JM, Curfs LM. Identifying effective methods for teaching sex education to individuals with intellectual disabilities: a systematic review. J Sex Res. 2015;52(4):412-32. doi: 10.1080/00224499.2014.919373. Epub 2014 Aug 1. PMID 25085114
- [Background] Jojo N, Nattala P, Seshadri S, Krishnakumar P, Thomas S. Knowledge of sexual abuse and resistance ability among children with intellectual disability. Child Abuse Negl. 2023 Feb;136:105985. doi: 10.1016/j.chiabu.2022.105985. Epub 2023 Jan 3. PMID 36603444